CLINICAL TRIAL: NCT05653505
Title: Safety and Efficacy of Remote Ischemic Conditioning Combined With Endovascular Stenting in Patients With Symptomatic Intracranial Atherosclerotic Stenosis
Brief Title: Remote Ischemic Conditioning Combined With Endovascular Stenting for Symptomatic Intracranial Atherosclerotic Stenosis
Status: Not yet recruiting | Type: Observational
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Chief Physician, Tianjin Huanhu Hospital
Other Study IDs: TJHH-2022-WM11
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Intracranial Arteriosclerosis; Ischemic Preconditioning; Endovascular Procedures
Keywords: Remote Ischemic Conditioning; Endovascular Stenting; Symptomatic Intracranial Atherosclerotic Stenosis
MeSH Terms: conditions — Intracranial Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular therapy: According to current guideline recommendations, patients enrolled in this cohort will receive standardized perioperative management, endovascular therapy, and postoperative medical therapy.
- Endovascular therapy+Remote ischemic conditioning: Patients enrolled in this cohort will receive the same treatment as those in the endovascular therapy alone cohort as well as additional remote ischemic conditioning treatment.
  Remote ischemic conditioning treatment protocol: RIC will be applied immediately after admission to the integrated neurovascular ward and the treatment continues until the patient is discharged, Once the patient is discharged, the choice of whether to continue RIC treatment depends on the patient's preference. RIC was induced through a standard blood pressure cuff placed around the non-paretic arm. The protocol includes 5 cycles of intermittent manually induced upper limb ischemia, alternating 5 minutes of inflation (20mmHg above systolic blood pressure), and 5 minutes of deflation twice a day.
  Interventions: Other: Remote Ischemic Conditioning

INTERVENTIONS:
Other: Remote Ischemic Conditioning — Remote ischaemic conditioning (RIC) refers to a process whereby periods of intermittent ischemia, typically via the cyclical application of a blood pressure cuff to a limb at above systolic pressure, confers systemic protection against ischemia in spatially distinct vascular territories.
  Groups: Endovascular therapy+Remote ischemic conditioning

SUMMARY:
The purpose of this registry is to evaluate the safety and efficacy of RIC for patients with symptomatic intracranial atherosclerotic stenosis (sICAS) undergoing endovascular therapy.

DETAILED DESCRIPTION:
Intracranial atherosclerotic stenosis (ICAS) is one of the leading causes of ischemic stroke, and its incidence varies widely among different ethnic groups. ICAS may represent approximately 10% of ischemic stroke in Caucasians and even be responsible for up to 50% in Chinese population. Recurrent stroke risks are as high as 23% 1 year after transient ischemic stroke (TIA) or stroke in patients with a stenosis of 70% or more. The Chinese IntraCranial AtheroSclerosis (CICAS) study indicated the prevalence of ICAS was 46.6%; Patients with ICAS had more severe stroke at admission and stayed longer in hospitals compared with those without intracranial stenosis. After 12 months, recurrent stroke occurred in 3.27% of patients with no stenosis, in 3.82% for those with 50% to 69% stenosis, in 5.16% for those with 70% to 99% stenosis, and in 7.27% for those with total occlusion.

Current guidelines recommend best medical treatment (BMM) for patients with sICAS, which contains antithrombotic therapy, management of vascular risk factor (diabetes, lipids, and especially hypertension) and patient behaviors modification (diet, exercise and smoking cessation). But, even with the intervention of BMM, the recurrence of ischemic stroke or transient ischemic attacks (TIAs) in patients with sICAS still cannot be reduced. Endovascular therapy with intracranial angioplasty and/or stenting holds great promise as a treatment for sICAS. A recent trial found that, compared with bare-metal stent, drug-eluting stent reduced the risks of In-stent restenosis and ischemic stroke recurrence in patients with sICAS. However, endovascular therapy for patients with sICAS is known to be associated with potentially serious complications such as cerebral hyper-perfusion syndrome, intracranial hemorrhage, embolism and In-stent restenosis, etc. Those are the main reasons that affect the effect of endovascular therapy, thus limiting its application and popularization to a great degree.

Remote Ischemic Conditioning (RIC) is one of the most potent neuroprotective approaches that can minimize neuronal damage by protecting against ischemia-reperfusion injury and promote neuronal recovery by stimulating endogenous protective mechanism through transiently occluding the blood supply to non-significant organs or tissues such as limbs. The investigators see a promising future for RIC in facilitating further clinical translation and application due to its unique features of safety, simplicity and non-invasiveness. In recent years, the safety and efficacy of RIC on stroke intervention has been confirmed by a series of basic and clinical researches, among which RIC in combination with adjuvant drug therapy for sICAS-induced ischemic stroke patient improve cerebral blood flow and reduce stroke recurrence. Since its safety and efficacy has been verified, RIC can also be used to reduce the risks of In-stent restenosis for patients with carotid stent implantation and has extensive application prospects for patients with severe acute ischemic stroke treated with endovascular thrombectomy.

There is not enough evidence as to provide any specific recommendation regarding the use of RIC in sICAS patients, But we speculate that RIC has a certain effect on preventing perioperative complications for patients with sICAS undergoing endovascular therapy. Therefore, we intend to conduct this prospective cohort study to shed light on the utility of this promising therapy.

This study prospectively collects data of patients with sICAS who receive endovascular therapy in the Comprehensive Neurovascular Ward of Tianjin Huanhu Hospital. Depending on their preference, patients enrolled in this registry will be divided into 2 groups, receiving either endovascular therapy alone or endovascular therapy plus RIC respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patient admitted from Jan. 1st 2023 to Jan. 1st 2025;
2. Age ≥ 18;
3. Intracranial atherosclerosis stenosis measured as ≥70% by digital subtraction angiography or by other noninvasive methods, such as transcranial doppler, computed tomography angiography, or magnetic resonance angiography;
4. A history of stroke/transient ischemic attack attributed to ICAS;
5. Verbal and written informed consent is provided at the time of admission by patients or their legally authorized representatives.

Exclusion Criteria:

1. Stenosis of other causes;
2. Prior ipsilateral stroke with residual deficits;
3. Uncontrolled hypertension (defined as systolic blood pressure ≥200 mm Hg despite medications at enrollment);
4. Peripheral vascular disease (especially subclavian arterial and upper limb artery stenosis or occlusion).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study prospectively collects data of patients with sICAS who receive endovascular therapy in the Comprehensive Neurovascular Ward of Tianjin Huanhu Hospital. Depending on their preference, patients enrolled in this registry will be divided into 2 groups, receiving either endovascular therapy alone or endovascular therapy plus RIC respectively.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The presence of ≥1 new brain lesions on DWI within 48 hours after endovascular stenting | 48 hours
  A new brain lesion was diagnosed if increased signal intensity was visible on DWI with correspondent decreased signal on apparent diffusion coefficient.
Incidence of clinical adverse events within 12 months after endovascular stenting | 12 months
  Clinical adverse events include ischemic stroke, TIA, acute myocardial infarction,hemorrhagic stroke, hyperperfusion syndrome, and death.

SECONDARY OUTCOMES:
Number of new brain lesions on DWI within 48 hours after endovascular stenting | 48 hours
  The number of new DWI lesions
The volume of new brain lesions on DWI within 48 hours after endovascular stenting | 48 hours
  The volume of single lesions, and volume of all lesions were measured on DWI.
National Institutes of Health Stroke Scale (NIHSS) scores at 12 months | 12 months
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Modified Rankin Scale (mRS) scores at 12 months | 12 months
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.functional disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Wei, PhD, Principal Investigator — Tianjin Huanhu Hospital
Locations (1):
- TianJinHH, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided